CLINICAL TRIAL: NCT03865407
Title: Uric Acid Reduction as a Novel Treatment for Pediatric Chronic Kidney Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: inability to achieve recruitment goals at a single center and given the current pandemic conditions
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20014698
Record Dates: First submitted 2019-03-05; First posted 2019-03-06 (Actual); Results first posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Hyperuricemia; Chronic Kidney Diseases
MeSH Terms: conditions — Hyperuricemia; Renal Insufficiency, Chronic | interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Allopurinol (Active Comparator): Allopurinol will be administered to this treatment arm group for 6 months. Participants will receive the lowest FDA recommended dose for weight, and will be titrated upwards to achieve the goal uric acid level of 3-5 mg/dL throughout the trial.
  Interventions: Drug: Allopurinol
- Standard of Care Control (No Intervention): The treatment arm will be compared to a standard of care arm.

INTERVENTIONS:
Drug: Allopurinol — Allopurinol dosed to target uric acid levels of 3-5 mg/dL.
  Arms: Allopurinol

SUMMARY:
Aim 1. To determine the effect of Allopurinol treatment on renal function (glomerular filtration rate, GFR) in pediatric chronic kidney disease (CKD) patients with high uric acid levels (hyperuricemia).

Aim 2. Establish whether Allopurinol treatment reduces Nlrp3 inflammasome and renal injury biomarkers.

DETAILED DESCRIPTION:
Uric acid levels often rise when kidney function declines. Historically, high uric acid has not been treated unless the uric acid crystallizes in the joint space and causes clinical gout disease, more typically seen in adults. However, new research has shown that high uric acid levels are associated with the development of hypertension, inflammation, and both acute and chronic kidney injury. Adult patients on renal dialysis who have hyperuricemia also have higher mortality rates. In several adult and in one pediatric clinical trial of uric acid lowering therapy (with Allopurinol or Febuxostat), treatment has demonstrated a slower rate of renal function decline and improved blood pressure compared to placebo. The pediatric trial was a 4-month placebo controlled trial of Allopurinol, and showed positive improvement in renal function and blood pressure, but did not adequately control for potential confounders in the outcome. Two known confounders that influence renal function (glomerular filitration rate, GFR) in pediatric CKD are race and glomerular or non-glomerular disease etiology. This study is designed to control for these confounders and establish whether Allopurinol for 6 months of treatment to a goal range of 3-5 mg/dL will improve renal function compared to standard of care. The secondary outcome is to determine whether blood pressure is affected by the treatment and the magnitude of change of serum uric acid. This study will also explore whether Allopurinol treatment alters activation of the Nlrp3 inflammasome or renal injury biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney Disease stage 1-5
* Hyperuricemic (UA >= 5.5 mg/dL)

Exclusion Criteria:

* Contraindication to Allopurinol
* Elevated baseline liver function tests
* Receiving acute or chronic dialysis
* Primary metabolic disorder
* Sickle cell disease
* Autosomal Dominant Polycystic Kidney Disease
* Cystinosis
* Bartter or Gitelman Disease
* Pregnant or nursing

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristin Kaspar, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Allopurinol | Standard of Care Control
Started | 10 | 7
Completed | 7 | 7
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Medical change caused patient to no longer meet inclusion/exclusion criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allopurinol | Standard of Care Control | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.29 (2.5) | 13.86 (2.61) | 14.07 (2.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: eGFR Change
Description: Change in Cys-C eGFR over time
Time Frame: The difference in Cystatin C eGFR between baseline and 6 months will be measured
Measure: Mean (Standard Deviation); unit: ml/min/1.73m^2
Arm/Group | Allopurinol | Standard of Care Control
Number analyzed (Participants) | 7 | 7
ml/min/1.73m^2 | 3.14 (3.716) | -0.29 (5.251)
Statistical Analysis 1: Comparison: Allopurinol vs Standard of Care Control; Test type: Superiority; p = 0.1839, t-test, 2 sided

2. Primary Outcome: eGFR Change
Description: Change in Creatinine eGFR over time
Time Frame: The difference in Creatinine eGFR between baseline and 6 months will be measured
Measure: Mean (Standard Deviation); unit: ml/min/1.73m^2
Arm/Group | Allopurinol | Standard of Care Control
Number analyzed (Participants) | 7 | 7
ml/min/1.73m^2 | 3.86 (7.798) | 0 (3.857)
Statistical Analysis 1: Comparison: Allopurinol vs Standard of Care Control; Test type: Superiority; p = 0.3036, t-test, 2 sided

3. Secondary Outcome: Serum Uric Acid Change
Description: Change in Serum Uric Acid
Time Frame: The difference in Serum Uric Acid between baseline and 6 months will be measured
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Allopurinol | Standard of Care Control
Number analyzed (Participants) | 7 | 7
mg/dl | -3.33 (0.996) | -0.46 (0.964)
Statistical Analysis 1: Comparison: Allopurinol vs Standard of Care Control; Test type: Superiority; p = 0.0001, t-test, 2 sided

4. Secondary Outcome: Systolic Blood Pressure
Description: Change in systolic blood pressure
Time Frame: The difference in clinic systolic blood pressure between baseline and 6 months will be measured
Population: Follow up blood pressure data was not collected from one participant in the treatment group
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Allopurinol | Standard of Care Control
Number analyzed (Participants) | 6 | 7
mmHg | -6.5 (13.126) | 2.29 (6.264)
Statistical Analysis 1: Comparison: Allopurinol vs Standard of Care Control; Test type: Superiority; p = 0.1421, t-test, 2 sided

5. Secondary Outcome: Diastolic Blood Pressure
Description: Change in diastolic blood pressure
Time Frame: The difference in clinic diastolic blood pressure between baseline and 6 months will be measured
Population: Follow up blood pressure data was not collected from one participant in the treatment group
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Allopurinol | Standard of Care Control
Number analyzed (Participants) | 6 | 7
mmHg | -7.33 (6.29) | 3.983 (7.543)
Statistical Analysis 1: Comparison: Allopurinol vs Standard of Care Control; Test type: Superiority; p = 0.0022, t-test, 2 sided

6. Other Pre Specified Outcome: Serum High Sensitivity C-reactive Protein (Hs-CRP)
Description: Compare the mean difference of serum hs-CRP from baseline to 6 months between groups
Time Frame: Serum hs-CRP will be measured at baseline and 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Allopurinol | Standard of Care Control
Number analyzed (Participants) | 7 | 7
mg/dL | 1.66 (3.724) | -7.64 (18.639)
Statistical Analysis 1: Comparison: Allopurinol vs Standard of Care Control; Test type: Superiority; p = 0.3032, t-test, 2 sided

7. Other Pre Specified Outcome: Interleukin 18
Description: Change in interleukin 18
Time Frame: Serum interleukin 18 will be measured at baseline, 3 months, and 6 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Serum Nlrp3
Description: Change in serum Nlrp3
Time Frame: Serum Nlrp3 will be measured at baseline, 3 months, and 6 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Urine Neutrophil Gelatinase-associated Lipocalin (NGAL)
Description: Change in urine NGAL
Time Frame: Urine NGAL will be measured at baseline, 3 months, and 6 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Urine Endothelin-1 (ET-1)
Description: Change in urine ET-1
Time Frame: Urine ET-1 will be measured at baseline, 3 months, and 6 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Urine Kidney Injury Molecule-1 (KIM-1)
Description: Change in urine KIM-1
Time Frame: Urine KIM-1 will be measured at baseline, 3 months, and 6 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Urine N-acetyl-Beta-D-Glucosaminidase (NAG)
Description: Change in urine NAG
Time Frame: Urine NAG will be measured at baseline, 3 months, and 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: Regular investigator assessment, regular laboratory testing
Arm/Group | Allopurinol | Standard of Care Control
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allopurinol (N=7) | Standard of Care Control (N=7)
Drug reaction with eosinophilia and systemic symptoms (DRESS) syndrome (Immune system disorders) | 1 (1) | 0 (0) — Patient in treatment intervention developed DRESS syndrome directly attributable to Allopurinol. Required renal replacement therapy, prolonged steroid taper and has partially recovered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT03865407/Prot_SAP_000.pdf